CLINICAL TRIAL: NCT03774004
Title: Association of Peripheral Atherosclerotic Burden With the Short-term and Long-term Outcome in Patients With Elective Myocardial Revascularisation
Brief Title: Plaque Burden Pre- Myocardial Revascularisation
Acronym: ByPlaque
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1098/2017
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective-observational, explorative single-centre cohort study aimed to examine the influence of the peripheral atherosclerotic plaque volume on short and long term morbidity and mortality in patient after coronary artery bypass grafting (CABG).

Atherosclerotic disease (IMT, plaque volume) will be measured with a ultrasound system (IMT measurements and 3D quantitative plaque volumetric). Hemodynamic and flow profiles of the internal thoracic arteries will be evaluated additionally with US. These parameters will be measured pre-CABG.

Morbidity will be evaluated using quality of life questionnaires (EQ-5D-3L, IPAQ). Major adverse cardiovascular events (MACE) will be the primary endpoint. The atherosclerotic burden will be compared with established risk scores (EuroSCORE, STS-Score, SYNTAX Score, FORECAST.

ELIGIBILITY:
Inclusion Criteria:

* pre CABG

Exclusion Criteria:

* no consent, prior carotid intervention

Ages: 30 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients, who are are listed for elective CABG at the Medical University Innsbruck will be screened and recruited.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Association of MACE rates with peripheral atherosclerotic volume | 5 years
Association of morbidity with peripheral atherosclerotic volume | 5 years
  Morbidity will be evaluated with quality of life assessment ("EQ-5D-3L", "IPAQ"

SECONDARY OUTCOMES:
Comparison of predictive value of peripheral atherosclerotic volume with established risk scores for cardiovascular operations and interventions | 1 year
  Risk scores include STS Score and Euro Score
Association of the duration of the operation with peripheral atherosclerotic volume | 30 days
Association of flow profiles of internal mammary artery with LIMA/RIMA graft patency rates | 5 years
Association of the aortic clamp time with peripheral atherosclerotic volume | 30 days
Association of the ICU stay with peripheral atherosclerotic volume | 30 days
Association of the hospitalization duration with peripheral atherosclerotic volume | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Marschang, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria